CLINICAL TRIAL: NCT05441046
Title: Phase I and Extended Clinical Study of Safety, Tolerability, and Pharmacokinetics of Injectable Genakumab Alone and Combination With Tislelizumab in the Treatment of Advanced Malignant Solid Tumors
Brief Title: Genakumab Alone and in Combination With Tislelizumab in Patients With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gensci048-ST-I
Record Dates: First submitted 2022-06-16; First posted 2022-07-01 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-05

CONDITIONS: Malignant Solid Tumors
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genakumab (Experimental): genakumab plus tislelizumab 200 mg
  Interventions: Drug: Genakumab

INTERVENTIONS:
Drug: Genakumab — genakumab plus tislelizumab 200 mg
  Other Names: Tislelizumab

SUMMARY:
This is a phase I, multicenter, open-label dose escalation and expansion study to evaluate genakumab alone and in combination with tislelizumab in adult patients with advanced solid malignancies.

DETAILED DESCRIPTION:
The study is divided into two parts:

Part I:

Part Ia: Two dose groups are planned, which are genakumab 200 mg, 300 mg. Genakumab is administered subcutaneously once every three weeks.

Part Ib: Three dose groups are planned, which are genakumab 100 mg plus tislelizumab 200 mg, genakumab 200 mg plus tislelizumab 200 mg, genakumab 300 mg plus tislelizumab 200 mg. Genakumab is administered subcutaneously once every three weeks. Tislelizumab is administered intravenously following genakumab on D1 of every cycle.

The study process of Part I includes the screening period (4 weeks), the observation period of dose-limiting toxicity (DLT) evaluation (defined as 3 weeks after first dosing), continuous dosing period (dosing once every 3 weeks until the discontinuation criteria are met), safety follow-up period after discontinuation (28±5 days after last dosing) and progression-free survival follow-up period after discontinuation (once every 6 weeks, until the progression-free survival follow-up endpoint).

Part II:

The sponsor and the investigator will choose one dose level as RP2D based on the totality of safety, PK, PD, and preliminary efficacy data from Part I. Additional 90 patients (30 patients for each cohort) will be treated at this dose level. The administration method is the same as that in Part I while without DLT observation.

ELIGIBILITY:
Inclusion Criteria:

Patients may be enrolled in the study only if they meet all of the following inclusion criteria:

1. Patients with advanced malignant tumors by histopathological diagnosis who do not have any acceptable standard treatments currently. Tumor types are specified as follows:

   Part I (Dose escalation): malignant solid tumors.

   Part II (Dose expansion):

   Cohort A: malignant solid tumors (excluding colorectal cancer and pancreatic cancer).

   Cohort B: colorectal cancer. Cohort C: pancreatic cancer.
2. Patients who have provided informed consent prior to initiation of any study-specific activities/procedures.
3. Age 18-75 years old.
4. Life expectancy ≥ 12 weeks.
5. Solid tumor with ≥ 1 measurable lesion that can be used to measure response according to RECIST v1.1. Index lesions must not be chosen from previously irradiated field unless there has been demonstrated disease progression in that lesion.
6. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Adequate organ function defined as follow:

   * Hematological (without need for hematopoietic growth factor or transfusion support within 14 days prior to screening) Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count (PLT) ≥ 75 x 109/L Hemoglobin (HGB) ≥ 90 g/L
   * Hepatic Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) OR ≤ 3 x ULN for patients with liver metastases or Gilbert syndrome Aspartate aminotransferase (AST) ≤ 2.5 x ULN OR ≤ 5 x ULN for patients with liver metastases Alanine aminotransferase (ALT) ≤ 2.5 x ULN OR ≤ 5 x ULN for patients with liver metastases
   * Renal Serum creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 45 mL/min (according to the Cockcroft-Gault equation)
   * Coagulation Activated thromboplastin time (aPTT) ≤ 1.5 x ULN International normalization ratio (INR) ≤ 1.5 x ULN If the patient is receiving anticoagulant therapy, the aPTT or INR must be in the therapeutic range of intended use of anticoagulants.
8. Female patients with the possibility of pregnancy: Agree to practice sexual abstinence or use effective methods of contraception from the time of signing the ICF until at least 6 months after the end of dosing. Male patients: Agree to practice abstinence or use effective contraception from the time of signing the ICF until at least 6 months after the end of dosing.

Patients who have recovered from the toxic effects of the last treatment (CTCAE ≤ grade 1, except for special circumstances such as "alopecia") before the first dosing.

Exclusion Criteria:

Patients with any of the following conditions may not be enrolled in the study:

1. Prior treatment with IL-1β-targeting agents.
2. Patients with previous severe allergic reactions to any investigational drugs or its components in this trial.
3. Previous or current other types of malignancy diagnosed within 3 years, except as follows: basal cell or squamous cell skin cancer that has been cured, any type of carcinoma in situ that has been cured.
4. Symptomatic central nervous system metastases. Patients with asymptomatic CNS metastases or patients who are radiologically and neurologically stable ≥ 2 weeks following CNS-directed therapy are eligible.
5. Patients who have received any of the following treatments within 4 weeks or within 5 half-lives prior to the first dosing (whichever is shorter):

   * Anti-tumor therapy (including chemotherapy, targeted therapy, immunotherapy, tumor artery embolization, and radiotherapy, excluding palliative radiotherapy);
   * Any biological agents targeting immune system (e.g., TNF blockers, anakinra, rituximab, abatacept or tocilizumab, etc);
   * Any live vaccines or live attenuated vaccines;
   * Any other investigational drugs or another interventional clinical study (except for the following: patients who participate in an observational, non-interventional clinical study, or are in the follow-up period of an interventional clinical study).
6. Major surgery or severe trauma within 4 weeks prior to the first dosing. Wounds and injuries must be fully recovered. Note: Video-assisted thoracoscopic surgery (VATS) and mediastinoscopy are not considered as major surgery. Patients who have received VATS or mediastinoscopy more than 2 weeks prior to the first dosing may be enrolled at the discretion of the investigator.
7. Patients who have a cardiovascular clinical condition or symptom including:

   * Unstable angina or myocardial infarction in the past 6 months;
   * Coronary artery bypass grafting (CABG) in the past 6 months;
   * Congestive heart failure (NYHA class 2);
   * Clinically significant malignant arrhythmia (e.g., persistent ventricular tachycardia, clinically significant second- or third-degree atrioventricular block without a pacemaker).
8. Uncontrolled diabetes or hypertension defined by the investigator.
9. History of interstitial lung disease.
10. Active or recurrent liver disease, including hepatitis B, hepatitis C, and liver cirrhosis.
11. Patients with active pulmonary tuberculosis found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection before enrollment (Patients who have received anti-tuberculosis treatment and further examinations confirm that there is no evidence of active infection are eligible.).
12. Patients with active infection requiring systematic treatment within 2 weeks prior to the first dosing (Patients with skin infection requiring only topical treatment are eligible.).
13. Patients with suspected or proven immunocompromised state, including:

    * Patients with evidence of Human Immunodeficiency Virus (HIV) infection;
    * Patients requiring systemic or local treatment with any immune modulating agent in doses with systemic effects e.g., high dose oral or intravenous steroids (> 10 mg/d prednisone or its equivalents) or high dose methotrexate (> 15 mg weekly). Topical, inhaled, local steroid use in doses that are not considered to cause systemic effects are permitted.
    * Patients with active or recurrent autoimmune disease, excluding: hypothyroidism with replacement therapy, skin disease without need for systemic treatment;
    * Patients with history of allogenic hematopoietic stem cell transplantation or organ transplantation (except corneal transplantation);
    * Patients with any other medical condition which in the opinion of the investigator places the patients at unacceptable risk for participation in immunomodulatory therapy.

Female patients who are pregnant or lactating, or have a positive pregnancy test result at baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicities (DLTs) | First cycle (21 days after first dose)
adverse events (AEs) adverse events (AEs) | through study completion, an average of 6 months
serious adverse events (SAEs) | through study completion, an average of 6 months
PK parameters of genakumab: bioavailability | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
PK parameters of genakumab: peak concentration (Cmax) | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
PK parameters of genakumab: area under time-concentration curve (AUC) | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
PK parameters of genakumab: t1/2 | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
PK parameters of genakumab: steady-state peak concentration | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
PK parameters of genakumab: steady-state trough concentration | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
PK parameters of genakumab: accumulation ratio | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months

SECONDARY OUTCOMES:
Pharmacodynamic: hsCRP | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
Pharmacodynamic: total IL-1β | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
Pharmacodynamic: free IL-1β | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
Pharmacodynamic: IL-6 | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
Pharmacodynamic: IL-8 | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months
Pharmacodynamic: TNF-α. | Cycle 1 day 1/day 2/day 3/day 4/day 6/day 8/day 15, Cycle 2 day 1, Cycle 3 day 1, Cycle 4 day 1/day 2/day 3/day 4/day 6/day 8/day 15, and day 1 of every following cycles (every cycle is 21 days) through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China